CLINICAL TRIAL: NCT06349226
Title: Development of New Diagnostic, Prognostic and Therapeutic Strategies in the Field of Degenerative Disc Disease: Identification of Biomarkers and Molecular Targets Involved in Discogenic Pain and Neuroinflammation
Brief Title: Identification of Biomarkers and Molecular Targets Involved on Intervertebral Disc Degeneration and Discogenic Pain
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: DISCOLAB
Record Dates: First submitted 2024-03-21; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Intervertebral Disc Degeneration; Discogenic Pain; Discogenic Disease
Keywords: intervertebral disc degeneration; discogenic pain; biomarkers; neuroinflammation; iperinnervation; sphingolipids; sphingosine-1 phosphate
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cells from human intervertebral disc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cell isolation from intervertebral disc tissue and biomarker investigation — metabolomic, cellular and molecular analysis on intervertebral disc derived cells and investigation of tissue neuroinflammatory and pain-related biomarkers

SUMMARY:
Low back pain, associated with intrinsic disorders of the spine, is a very frequent clinical condition that is accompanied by high morbidity with effects both on psychosocial aspects, and health care system. It occurs in approximately 80% of the population throughout their lives. Most low back pain is associated with intervertebral disc degeneration (IDD) associated with neuroinflammation and pain. In this context, the study of sphingolipid metabolism can play an important role in the identification of new molecules responsible for the degenerative process. Sphingolipids, in fact, are a class of molecules that are implicated in multiple signal pathways, such as proliferation, degradation of the extracellular matrix, inflammatory state, apoptosis and migration. In particular, sphingosine-1-phosphate (S1P), an intermediate of sphingolipid metabolism, acts as a pro-inflammatory mediator, predominantly in the extracellular environment, regulating important cellular properties related to inflammatory potential and pain. The objective of this study is to characterize the degenerative process in cells isolated from degenerated human intervertebral discs from both at cellular and molecular levels in order to identify new targets implicated in degenerative processes, including sphingolipid signaling pathway.

DETAILED DESCRIPTION:
Low back pain (LBP) is a serious public health problem and has been identified as the most widespread cause of disability worldwide by the 2013 Global Burden of Disease Study. It is estimated that in the Western world the annual incidence of acute low back pain is 5% in adults and that the lifetime prevalence is 80%. Although different anatomical structures can be implicated in the generation of LBP, in many cases this is associated with the degeneration of the intervertebral disc (IVD). IVD degeneration (IDD) represents a chronic age-related process, characterized by a progressive reduction in the content of proteoglycans and water in the nucleus pulposus (NP) with the subsequent loss of the ability of the disc to respond to compressive forces with the possible appearance of instability. Furthermore, this degenerative process is accompanied by the development of a highly inflammatory microenvironment which contributes to exacerbating the degenerative process, leading to the progressive structural failure of the disc itself and in most cases, to pain. From these premises, arises the need to better investigate all the cell-mediated mechanisms underlying IDD, to identify and develop new therapies aimed at recovering the IVD and reducing pain.

In this context, sphingolipids, a class of molecules responsible for multiple signal pathways such as proliferation, migration, apoptosis and angiogenesis, appear to play a key role in exacerbating the inflammatory process and degradation of the extracellular matrix in conditions of IDD. Sphingosine-1-phosphate (S1P) is an intermediate of sphingolipid metabolism, formed from sphingosine through the action of sphingosine kinases (SphK1, SphK2). Increasing evidence suggests that S1P acts as a pro-inflammatory signal, predominantly in the extracellular environment, regulating important cellular properties correlated with the inflammatory potential on chondrocyte-like cells. It has been reported that an alteration in the production and secretion of these molecules is capable of increasing the inflammatory and degenerative condition in various pathologies related to neuroinflammation and pain. The aim of the project is to define new disease biomarkers and characterize the degenerative process in cells isolated from degenerated human intervertebral discs from both at cellular and molecular levels in order to identify new targets implicated in degenerative processes, including sphingolipid signaling pathway. Secondary objective is the analysis of the effectiveness of the modulation of sphingolipid metabolism and the in vitro testing of molecules with therapeutic potential.

A greater understanding of the events implicated in the pathogenesis of IDD both at macroscopic and microscopic levels, is of fundamental importance for the development of new diagnostic tools, to be combined with current therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with disc degeneration for spondylolisthesis, herniated intervertebral disc, and other causes of disc degeneration

Exclusion Criteria:

* Spinal infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent the surgery of discectomy for the degenerative disc.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2025-05-21 (Estimated); Study Completion 2025-05-21 (Estimated)

PRIMARY OUTCOMES:
Characterization of degenerated intervertebral disc cells | through study completion, an average of 3 years
  Determination of a panel of inflammatory and degenerated markers related to components of the extracellular matrix and mediators linked to inflammatory/degenerative processes, hyperinnervation and sphingolipid metabolism.

SECONDARY OUTCOMES:
Development of cellular model platform | through study completion, an average of 3 years
  Creation of a cellular platform based on patient-derived intervertebral disc cells; assessment of inflammatory and degenerative markers linked to alteration of sphingolipid metabolism; determination of a panel of inflammatory cytokines related to degenerative process, neuro-inflammation and pain; evaluation of prognostic and predictive markers related to disc degeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Locatelli, MD, PhD, Study Director — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Neurosurgery Unit; Mauro Pluderi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Neurosurgery Unit; Giovanni Marfia, MD, PhD, Study Chair — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Neurosurgery Unit, Istituto di Medicina Aerospaziale di Milano, CeMATA - Aeronautica Militare
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Result] Marfia G, Guarnaccia L, Navone SE, Ampollini A, Balsamo M, Benelli F, Gaudino C, Garzia E, Fratocchi C, Di Murro C, Ligarotti GK, Campanella C, Landolfi A, Perelli P, Locatelli M, Ciniglio Appiani G. Microgravity and the intervertebral disc: The impact of space conditions on the biomechanics of the spine. Front Physiol. 2023 Mar 14;14:1124991. doi: 10.3389/fphys.2023.1124991. eCollection 2023. PMID 36998982
- [Result] Navone SE, Campanella R, Guarnaccia L, Ouellet JA, Locatelli M, Cordiglieri C, Gualtierotti R, Gaudino C, Ciniglio Appiani G, Luzzi S, Borsa S, Rampini P, Pluderi M, Haglund L, Riboni L, Alini M, Marfia G. Inflammatory interactions between degenerated intervertebral discs and microglia: Implication of sphingosine-1-phosphate signaling. J Orthop Res. 2021 Jul;39(7):1479-1495. doi: 10.1002/jor.24827. Epub 2020 Aug 24. PMID 32779775
- [Result] Navone SE, Peroglio M, Guarnaccia L, Beretta M, Grad S, Paroni M, Cordiglieri C, Locatelli M, Pluderi M, Rampini P, Campanella R, Alini M, Marfia G. Mechanical loading of intervertebral disc modulates microglia proliferation, activation, and chemotaxis. Osteoarthritis Cartilage. 2018 Jul;26(7):978-987. doi: 10.1016/j.joca.2018.04.013. Epub 2018 May 1. PMID 29723636
- [Result] Navone SE, Marfia G, Giannoni A, Beretta M, Guarnaccia L, Gualtierotti R, Nicoli D, Rampini P, Campanella R. Inflammatory mediators and signalling pathways controlling intervertebral disc degeneration. Histol Histopathol. 2017 Jun;32(6):523-542. doi: 10.14670/HH-11-846. Epub 2016 Nov 16. PMID 27848245
- [Result] Marfia G, Campanella R, Navone SE, Zucca I, Scotti A, Figini M, Di Vito C, Alessandri G, Riboni L, Parati E. Potential use of human adipose mesenchymal stromal cells for intervertebral disc regeneration: a preliminary study on biglycan-deficient murine model of chronic disc degeneration. Arthritis Res Ther. 2014 Oct 8;16(5):457. doi: 10.1186/s13075-014-0457-5. PMID 25293819
- [Result] Marfia G, Navone SE, Di Vito C, Tabano S, Giammattei L, Di Cristofori A, Gualtierotti R, Tremolada C, Zavanone M, Caroli M, Torchia F, Miozzo M, Rampini P, Riboni L, Campanella R. Gene expression profile analysis of human mesenchymal stem cells from herniated and degenerated intervertebral discs reveals different expression of osteopontin. Stem Cells Dev. 2015 Feb 1;24(3):320-8. doi: 10.1089/scd.2014.0282. Epub 2014 Oct 29. PMID 25203751
- See also: website Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico — http://www.policlinico.mi.it/reparti/40/neurochirurgia